CLINICAL TRIAL: NCT02490059
Title: Ultrathin Bronchoscopy for Solitary Pulmonary Nodules: A Randomised Pilot Trial
Brief Title: Ultrathin Bronchoscopy for Solitary Pulmonary Nodules
Acronym: Babyscope
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: University of Stellenbosch (Other)
Responsible Party: Principal Investigator, Daniel Franzen, Medical Doctor, University of Zurich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2000-C094
Record Dates: First submitted 2015-06-25; First posted 2015-07-03 (Estimated); Last update posted 2015-07-03 (Estimated); Status verified 2015-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard size bronchoscopy (Active Comparator): ll procedures were started using SB with an external diameter of 5.0-6.0 mm with a biopsy channel of 2.2-2.8 mm (models Olympus BF-30 and BF-1T160, Olympus, Tokyo, Japan). If during SB the lesion was endoscopically visible the bronchoscopy was continued as standard diagnostic procedure and the patients were excluded from the analysis. Only if no tumour was visible during complete inspection of the bronchial tree using the SB, a participant was randomised by opening a numbered sealed opaque envelope. Randomisation was performed using sequentially numbered (1-40) sealed opaque envelopes (block randomisation: block size 4). For subjects allocated to the SB group, the examination was immediately continued with the same SB bronchoscope.
  Interventions: Other: bronchoscopy
- Ultrahin bronchoscopy (Experimental): For subjects randomised to UB, the instrument was changed immediately to an Olympus BF-XP 40 ultrathin bronchoscope with an outer diameter of 2.8 mm and a working channel 1.2 mm during the same bronchoscopy session.
  Interventions: Other: bronchoscopy

INTERVENTIONS:
Other: bronchoscopy — Bronchoscopy for diagnosis of pulmonary nodules

SUMMARY:
The evaluation of solitary pulmonary nodules (SPN) requires a balance between procedure-related morbidity and diagnostic yield, particularly in areas where tuberculosis is endemic. Data on ultrathin bronchoscopy (UB) for this purpose is limited. In this prospective randomised trial we compared diagnostic yield and adverse events of UB with standard-size bronchoscopy (SB) in a cohort of patients with SPN located beyond the visible range of SB.

DETAILED DESCRIPTION:
The present prospective single-centre randomised pilot study was performed at Tygerberg Academic Hospital, a tertiary university hospital in Cape Town, South Africa, with a referral drainage area of 1.5 million people and tuberculosis notification rate of up to 1'000/100'000 persons per year when the study was performed. Between November 2000 and November 2003 all patients referred to the lung unit with single pulmonary lesion ≤ 6 cm in diameter on chest computed tomography (CT) were included. SPN was defined as a single and circumscribed pulmonary lesion with a diameter ≤ 6.0 cm, surrounded by aerated lung tissue, and without evidence of atelectasis, pneumonitis, or cavity on CT scan. Location and maximal diameter of all SPNs were recorded from the chest CT prior to enrolment of patients. Inclusion criteria were a previous cytological and microbiological negative sputum examination, absence of enlarged mediastinal or hilar lymph nodes on chest CT scan, and informed consent obtained before start of the procedure. Exclusion criteria were SPN with lesion size unchanged over two years, inability to undergo bronchoscopy or thoracotomy, and pregnancy. Participants with consent for participation in the study in whom the lesion was found to be visible on SB were then not randomised and not considered part of the study population. Written informed consent was obtained from all patients before inclusion in the study.

ELIGIBILITY:
Inclusion Criteria:

* Pulmonary nodule on a recent CT
* non-visible on standard-size bronchoscopy

Exclusion Criteria:

* missing informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2000-11; Primary Completion 2003-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Sensitivity | 2 years
  Sensitivity of the diagnosis of malignancy. Biopsy specimens obtained by bronchoscopy were compared with the diagnosis made by surgical resection or CT-guided trans-thoracic needle aspiration if applicable. Efforts were made to obtain confirmatory histological diagnosis for all patients. Alternatively, when invasive diagnosis was not feasible or appropriate (as assessed by a multidisciplinary tumour board) radiological follow-up examinations were performed over two years.

SECONDARY OUTCOMES:
Diagnostic yield | 2 years
  Diagnostic yield of UB compared to SB. Biopsy specimens obtained by bronchoscopy were compared with the diagnosis made by surgical resection or CT-guided trans-thoracic needle aspiration if applicable. Efforts were made to obtain confirmatory histological diagnosis for all patients. Alternatively, when invasive diagnosis was not feasible or appropriate (as assessed by a multidisciplinary tumour board) radiological follow-up examinations were performed over two years.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Franzen, MD, Principal Investigator — University of Zurich
Locations (1):
- University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Derived] Franzen D, Diacon AH, Freitag L, Schubert PT, Wright CA, Schuurmans MM. Ultrathin bronchoscopy for solitary pulmonary lesions in a region endemic for tuberculosis: a randomised pilot trial. BMC Pulm Med. 2016 Apr 27;16(1):62. doi: 10.1186/s12890-016-0225-1. PMID 27117455